CLINICAL TRIAL: NCT02848430
Title: Hop Botanical Dietary Supplements - Metabolism and Safety in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Richard B van Breemen, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0651
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Food-Drug Interactions
Keywords: Humulus lupulus
MeSH Terms: interventions — ALPL protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Humulus lupulus (Experimental): Spent hop extract; 2 gelatin capsules (59.5 mg extract) per day for 14 days
  Interventions: Dietary Supplement: Humulus lupulus

INTERVENTIONS:
Dietary Supplement: Humulus lupulus — Extract of spent hops standardized to xanthohumol, isoxanthohumol, 6-prenylnaringenin, and 8-prenylnaringenin
  Other Names: hops

SUMMARY:
Human safety studies were carried out to test whether hop botanical dietary supplements used by peri- and post-menopausal women are safe to use with Food and Drug Administration (FDA)-approved drugs. To test this, a hop dietary supplement (previously tested in women at the University of Illinois at Chicago without any harmful effects) was given with four selected FDA-approved drugs to determine if the hop supplement can increase or decrease how these medications are absorbed, metabolized and excreted by the human body. Preclinical studies had predicted that the hop supplement might affect the metabolism or break down of these probe drugs.

DETAILED DESCRIPTION:
At the start of a study, subjects were administered low doses of a mixture of four FDA-approved drugs (caffeine, tolbutamide, dextromethorphan, and alprazolam), and serial blood samples were drawn and analyzed for the concentration of each drug over time. Afterwards, participants consumed the hop dietary supplement twice daily for 14 days to allow for potential inhibition or induction of drug metabolizing enzymes and transporters. Thereafter, the same drugs were taken again to obtain a second measure of drug concentrations in blood over time. Changes in the concentration-time curve values for each probe drug obtained before and after ingestion of the supplement would indicate that metabolism of the probe drugs is impacted by the hop dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* healthy peri- and post-menopausal women ages 40 - 79
* non-smokers
* no-significant medical conditions as assessed by subject-reported medical history, physical examination and blood and urine chemistry screens
* no medical condition that requires chronic use of medication

Exclusion Criteria:

* known allergies or hypersensitivity to caffeine, dextromethorphan, sulfonylureas (tolbutamide), benzodiazepines, red clover, licorice, or hops
* positive pregnancy test
* use of hormone therapy within 8 weeks of study initiation for oral agents, 4 weeks for transdermal or other topical agents
* use of caffeine products 7 days before study participation or during the study
* use of citrus products 7 days before study participation or during the study
* use of other prescription (with the exception of the Mirena® IUD) or non-prescription medicines within the 2 weeks prior to study initiation or during the study
* chronic diseases, such as inflammatory bowel disease, that could alter the absorption or metabolism of the probe substrates
* unwillingness to comply with study requirements
* current participation in another clinical trial
* CYP2D6 deficiency based on phenotyping at screening
* smoker
* hops intake (whether as a botanical dietary supplement or beer) within the previous two weeks and during the study
* use of any dietary supplements within the last 2 weeks prior to study initiation and during the study
* obesity (defined as >33 BMI)
* alcohol or drug abuse
* chronic diseases such as inflammatory bowel disease or diabetes

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention were used to calculate area under the (extrapolated) concentration-time curve to determine any changes compared to pre-intervention.

SECONDARY OUTCOMES:
Apparent Clearance | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention were used to calculate area under the (extrapolated) concentration-time curve to determine any changes compared to pre-intervention.
Peak Concentration | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention were used to calculate peak concentration of probe drug to determine any changes compared to pre-intervention.
Time for Peak Concentration | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention were used to calculate time for peak concentration of probe drug to determine any changes compared to pre-intervention.
Drug Half-life | baseline and 14 days
  Concentration of probe drugs from blood draws during the 14-day intervention were used to calculate half-life of probe drug to determine any changes compared to pre-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B van Breemen, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Breemen RB, Yuan Y, Banuvar S, Shulman LP, Qiu X, Alvarenga RF, Chen SN, Dietz BM, Bolton JL, Pauli GF, Krause E, Viana M, Nikolic D. Pharmacokinetics of prenylated hop phenols in women following oral administration of a standardized extract of hops. Mol Nutr Food Res. 2014 Oct;58(10):1962-9. doi: 10.1002/mnfr.201400245. Epub 2014 Sep 16. PMID 25045111
- [Result] van Breemen RB, Chen L, Tonsing-Carter A, Banuvar S, Barengolts E, Viana M, Chen SN, Pauli GF, Bolton JL. Pharmacokinetic Interactions of a Hop Dietary Supplement with Drug Metabolism in Perimenopausal and Postmenopausal Women. J Agric Food Chem. 2020 May 6;68(18):5212-5220. doi: 10.1021/acs.jafc.0c01077. Epub 2020 Apr 24. PMID 32285669
- See also: University of Illinois at Chicago / National Institutes of Health Center for Botanical Dietary Supplements — https://pharmacy.uic.edu/research/botanical-dietary-supplements